CLINICAL TRIAL: NCT07378761
Title: Efficacy of Ursodeoxycholic Acid Versus Corticosteroids for the Treatment of Cholestatic Hepatitis Secondary to Immunotherapy: A Multicenter, Controlled, Randomized, Open Trial
Brief Title: Comparing UDCA and Corticosteroids in Immunotherapy Induced Cholestatic Hepatitis
Acronym: CHILURSO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL24_0328; 2025-521317-50-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Immune-Mediated Cholestasis
Keywords: DILI; Immune checkpoint inhibitors; Cancer; Cholestatic hepatitis
MeSH Terms: conditions — Neoplasms | interventions — Ursodeoxycholic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients randomized to the experimental arm will receive ursodeoxycholic acid (UDCA) as initial treatment for hepatitis. After evaluation of the primary endpoint at Day 21, UDCA treatment will be continued for a total duration of 6 months. In case of lack of response to UDCA, patients will continue UDCA and will additionally receive corticosteroids which represent the reference treatment.
  Interventions: Drug: UDCA (Ursodeoxycholic acid)
- Control arm (Active Comparator): Patients randomized to the control arm will receive the reference treatment, corticosteroids. Corticosteroids will be given at a dose of 0.5-1 mg/kg/day for 21 days, followed by tapering in weekly steps of 10 mg until treatment discontinuation. At Day 21, in case of lack of treatment response, defined as no decrease of alkaline phosphatase and/or gamma-glutamyl transferase levels of at least 25% compared with baseline, corticosteroid tapering will continue, and ursodeoxycholic acid (UDCA) will be added at a dose of 13-15 mg/kg/day.
  Interventions: Drug: Corticosteroids (Reference Treatment)

INTERVENTIONS:
Drug: UDCA (Ursodeoxycholic acid) — Ursodeoxycholic acid (UDCA) will be administered orally at an initial dose of 13-15 mg/kg/day, divided into two daily doses. After assessment of the primary endpoint at Day 21, UDCA will be continued for a total treatment duration of 6 months. In case of absence of treatment response, defined as no decrease of alkaline phosphatase and/or gamma-glutamyl transferase levels of at least 25% compared with baseline, corticosteroids which represent the reference treatment, will be added at a dose of 0.5-1 mg/kg.
  Arms: Experimental arm
Drug: Corticosteroids (Reference Treatment) — Corticosteroids will be administered orally at a dose of 0.5-1 mg/kg/day for 21 days, followed by a tapering schedule of 10 mg per week until treatment discontinuation. At Day 21, if there is no adequate response (defined as less than 25% decrease in alkaline phosphatase and/or gamma-glutamyl transferase from baseline), the corticosteroid taper will continue and ursodeoxycholic acid (UDCA) will be added at a dose of 13-15 mg/kg/day.
  Arms: Control arm

SUMMARY:
The clinical trial aims to compare the effectiveness of ursodeoxycholic acid (UDCA) to corticosteroids in treating cholestatic hepatitis induced by immune checkpoint inhibitors (ICIs) over a 21-day period.

The trial presents a detailed scientific justification for comparing UDCA to corticosteroids, describing the treatment and detailing the follow-up procedures. It hypothesizes that UDCA could be superior to corticosteroids for treating ICI-related cholestatic hepatitis, based on its established use in primary biliary cholangitis and a favorable tolerance profile compared to corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Any type of cancer except hepatocellular or cholangiocarcinoma
* At least one ICI injection
* Cholestatic hepatitis Grade CTC-AE 3 or 4

Exclusion Criteria:

* Ongoing corticosteroids treatment
* Other causes of hepatitis
* Cirrhosis
* ICI for hepatocellular carcinoma or cholangiocarcinoma
* Biliary obstruction
* Medical contraindication to corticosteroids or UDCA
* Mixed or hepatocellular hepatitis
* Total bilirubin > 1,5 ULN, Prothrombin rate < 70%
* Medical contraindication to MRI or liver biopsy
* Oher serious side effects requiring corticosteroids
* Pregnant and breast-feeding patients
* Patients under articles L1121-5 to 8 of the public health code
* Lack of informed consent
* Patients not affiliated with French social security system
* Patients uncapable of understanding french

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Improvement of at least 25% in liver function tests on day 21 after randomization | 21 days after randomization
  The rate of patients showing an improvement of at least 25% in liver function tests (alkaline phosphatase and/or gamma-GT) on Day 21 after randomization.

SECONDARY OUTCOMES:
Rate of Hepatitis Resolution at 6 Months | 6 Months after randomization
  Rate of patients with resolution of hepatitis, defined as hepatitis grade ≤ 1 according to the current National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), at 6 months after randomization.
Time to Hepatitis Resolution | From Randomization to end of follow-up at 12 months
  Time to hepatitis resolution, defined as the time from the date of randomization to the date of hepatitis resolution (grade ≤ 1). Hepatitis severity will be graded according to the current National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Tolerance to UDCA and/or Corticosteroids | From treatment initiation following the randomization to end of follow-up at 12 months
  Tolerance to ursodeoxycholic acid (UDCA) and/or corticosteroids will be evaluated through the assessment of adverse events. Adverse events will be collected throughout the study and graded according to the current National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Resumption of immunotherapy | Within 12 months after randomization
  Rate of patients in whom resumption of immunotherapy was possible after hepatitis within 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Meunier, Principal Investigator — University Hospital, Montpellier
Locations (6):
- France (6):
  - CHU Bordeaux, Bordeaux
  - HCL Croix Rousse, Lyon
  - CHU Montpellier, Montpellier
  - APHP Paul Brousse, Paris
  - CHU Poitiers, Poitiers
  - CHU Toulouse, Toulouse